CLINICAL TRIAL: NCT06838923
Title: Effects of Light vs. Heavy Paraffin Oil on Embryo Culture in IVF: A Prospective Study on Development and Pregnancy Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hung Vuong Hospital (Other)
Responsible Party: Principal Investigator, Thi Thanh Thuy Tran, MD, Principal Investigator, Hung Vuong Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS/HV/24/25
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Embryo Development; Blastocyst IVF; Pregnancy Rates; IVF; Embryo Culture Media
Keywords: heavy/light paraffin oil for embryo culture

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment model, where participants undergoing in vitro fertilization (IVF) are randomly assigned to one of two groups. In the light paraffin oil group, embryos are cultured under conditions using light paraffin oil, while in the heavy paraffin oil group, embryos are cultured using heavy paraffin oil. The study aims to compare the effects of these two oil types on embryo development and pregnancy outcomes.
  Participants remain in their assigned group throughout the study without crossover between interventions. Key outcomes, including embryo development, blastocyst formation rate, and pregnancy rate, will be evaluated to determine which oil type provides optimal conditions for embryo culture in IVF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light Paraffin Oil Group (Experimental): Embryos are cultured under light paraffin oil conditions.
  Interventions: Combination Product: Light Paraffin Oil
- Heavy Paraffin Oil Group (Experimental): Embryos are cultured under heavy paraffin oil conditions. Thus, the Number of Arms = 2.
  Interventions: Combination Product: Heavy Paraffin Oil

INTERVENTIONS:
Combination Product: Light Paraffin Oil — Embryos in this group will be cultured under conditions using light paraffin oil as an overlay in in vitro fertilization (IVF). The oil serves to protect the culture media from evaporation and temperature fluctuations. Key outcomes, including embryo development, blastocyst formation rate, and pregnancy rate, will be assessed.
  Arms: Light Paraffin Oil Group
Combination Product: Heavy Paraffin Oil — Embryos in this group will be cultured under conditions using heavy paraffin oil as an overlay in in vitro fertilization (IVF). This study aims to compare the effects of heavy paraffin oil to light paraffin oil in embryo culture, assessing embryo development, blastocyst formation, and pregnancy rates.
  Arms: Heavy Paraffin Oil Group

SUMMARY:
This prospective study aims to compare the effects of light and heavy paraffin oil in embryo culture during in vitro fertilization (IVF). Paraffin oil is commonly used in IVF laboratories to protect embryo culture media from evaporation and temperature fluctuations. However, the impact of different oil viscosities on embryo development and pregnancy outcomes remains unclear.

Participants undergoing IVF treatment will have their embryos cultured under either light or heavy paraffin oil conditions. The study will evaluate key outcomes, including embryo development, blastocyst formation rates, and pregnancy rates. Findings from this research may help optimize embryo culture conditions, potentially improving IVF success rates and guiding best laboratory practices.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing in vitro fertilization (IVF) treatment with planned embryo culture.
* Patients with normal ovarian function or undergoing ovarian stimulation for IVF.
* Willingness to participate and provide informed consent.

Exclusion Criteria:

* Presence of severe uterine abnormalities (e.g., congenital malformations, Asherman's syndrome).
* History of recurrent implantation failure (≥3 unsuccessful IVF attempts).
* Poor ovarian response (e.g., ≤3 oocytes retrieved in a previous IVF cycle).
* Presence of severe male factor infertility, requiring testicular sperm extraction (TESE) or micro-TESE.
* Use of pre-implantation genetic testing (PGT) for embryo selection.
* Known autoimmune disorders or uncontrolled chronic conditions (e.g., diabetes, thyroid disorders) that may affect pregnancy outcomes.
* Participation in another clinical trial that may interfere with study outcomes.
* Donor cycles or surrogacy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 818 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Fertilization Rate | 16-20 hours post-insemination
  The proportion of oocytes that successfully undergo fertilization after insemination, as determined by the presence of two pronuclei (2PN) at the appropriate time post-fertilization.
Cleavage Rate | 48 hours post-fertilization
  The proportion of fertilized oocytes that progress to cleavage-stage embryos, assessed by the number of embryos that reach at least the two-cell stage within 48 hours after fertilization.
Blastocyst Formation Rate | 5-6 days post-fertilization
  The proportion of embryos that successfully develop into blastocysts by Day 5 or Day 6 of culture, assessed based on morphological grading criteria.

SECONDARY OUTCOMES:
Positive Beta-hCG | 14 days post-embryo transfer
  The proportion of participants achieving a positive serum beta-hCG test, indicating biochemical pregnancy, measured approximately two weeks after embryo transfer.
Implantation Rate | 4-5 weeks post-embryo transfer
  The proportion of transferred embryos that successfully implant in the uterus, determined by the presence of a gestational sac on ultrasound.
Clinical Pregnancy Rate | 6-7 weeks post-embryo transfer
  The proportion of participants with ultrasound-confirmed pregnancy, defined by the presence of a gestational sac with fetal heartbeat.
Ongoing Pregnancy Rate | 12 weeks post-embryo transfer
  The proportion of participants with a viable pregnancy continuing beyond the first trimester (≥12 weeks of gestation).
Live Birth Rate | At delivery (up to ~40 weeks of gestation)
  The proportion of participants who achieve a live birth, defined as the delivery of a viable infant at ≥24 weeks of gestation.
Pregnancy Loss Rate | From positive beta-hCG until delivery
  The proportion of participants experiencing pregnancy loss at any stage

CONTACTS AND LOCATIONS:
Locations (1):
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding patient confidentiality and privacy, in accordance with ethical guidelines and regulatory requirements for fertility treatment studies. Additionally, since this study involves sensitive reproductive health data, data sharing is restricted to aggregate-level results to protect participant anonymity.
  However, summary findings and statistical analyses will be made available through peer-reviewed publications and conference presentations to ensure transparency and contribution to scientific knowledge.